CLINICAL TRIAL: NCT01676220
Title: 6-Month, Multicenter, Randomized, Open-label, Parallel-group Study Comparing the Efficacy and Safety of a New Formulation of Insulin Glargine and Lantus® in Insulin-Naïve Patients With Type 2 Diabetes Mellitus Not Adequately Controlled With Non-Insulin Antihyperglycemic Drugs With a 6-month Safety Extension Period
Brief Title: Comparison of a New Formulation of Insulin Glargine With Lantus in Patients With Type 2 Diabetes on Non-insulin Antidiabetic Therapy
Acronym: EDITION III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC12347; 2012-000146-35 (EudraCT Number); U1111-1124-5261 (Other: UTN)
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOE901-U300 (Experimental)
  Interventions: Drug: HOE901-U300 (new formulation of insulin glargine)
- Lantus (Active Comparator)
  Interventions: Drug: Lantus (insulin glargine)

INTERVENTIONS:
Drug: HOE901-U300 (new formulation of insulin glargine) — HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily (evening) for 12 months on top of non-insulin antihyperglycemic drug(s). Dose titration seeking fasting plasma glucose 4.4-5.6 millimole per liter (mmol/L) (80 - 100 milligram per deciliter [mg/dL]).
  Arms: HOE901-U300
Drug: Lantus (insulin glargine) — Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily (evening) for 12 months on top of non-insulin antihyperglycemic drug(s). Dose titration seeking fasting plasma glucose 4.4-5.6 mmol/L (80 - 100 mg/dL).
  Other Names: Lantus
  Arms: Lantus

SUMMARY:
Primary Objective:

To compare the efficacy of a new formulation of insulin glargine and Lantus in terms of change of HbA1c from baseline to endpoint (scheduled at Month 6, Week 26) in participants with type 2 diabetes mellitus

Secondary Objectives:

To compare a new formulation of insulin glargine and Lantus in terms of:

- occurrence of nocturnal hypoglycemia

DETAILED DESCRIPTION:
The maximum study duration was up to approximately 54 weeks per participant, consisting of:

* Up to 2 week screening period; it can be exceptionally extended of up to one additional week
* 6-month comparative efficacy and safety treatment period
* 6-month comparative safety extension period
* 2-day post-treatment safety follow-up period

ELIGIBILITY:
Inclusion criteria :

* Adult participants with type 2 diabetes mellitus inadequately controlled with non-insulin antihyperglycemic drug(s);
* Signed written informed consent.

Exclusion criteria:

* HbA1c less than (<) 7.0% (< 53 millimole per mole [mmol/mol]) or greater than (>) 11% (> 97 mmol/mol)
* History of type 2 diabetes mellitus for less than 1 year before screening
* Less than 6 months before screening with non-insulin antihyperglycemic treatment
* Change in dose of non-insulin antihyperglycemic treatment in the last 3 month before screening
* Initiation of new glucose-lowering medications and/or weight loss drug in the last 3 months before screening visit and/or initiation of Glucagon-like peptide-1 (GLP-1) receptor agonist in the last 6 months before screening visit
* Participants receiving only non-insulin antihyperglycemic drugs not approved for combination with insulin according to local labeling/local treatment guidelines and/or sulfonylurea or glinide (Note: non-insulin antihyperglycemic drugs not approved for combination with insulin, sulfonylurea and glinide are to be discontinued at baseline)
* Current or previous insulin use except for a maximum of 8 consecutive days (for example, acute illness, surgery) during the last year prior to screening
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require treatment (for example, laser, surgical treatment or injectable drugs) during the study period

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 878 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (217):
- United States (117):
  - Investigational Site Number 840324, Montgomery, Alabama
  - Investigational Site Number 840273, Chandler, Arizona
  - Investigational Site Number 840217, Mesa, Arizona
  - Investigational Site Number 840220, Peoria, Arizona
  - Investigational Site Number 840211, Phoenix, Arizona
  - Investigational Site Number 840207, Phoenix, Arizona
  - Investigational Site Number 840264, Tempe, Arizona
  - Investigational Site Number 840234, Tempe, Arizona
  - Investigational Site Number 840304, Little Rock, Arkansas
  - Investigational Site Number 840347, Bell Gardens, California
  - Investigational Site Number 840244, Escondido, California
  - Investigational Site Number 840257, Fresno, California
  - Investigational Site Number 840213, Greenbrae, California
  - Investigational Site Number 840267, Huntington Beach, California
  - Investigational Site Number 840230, La Jolla, California
  - Investigational Site Number 840235, La Mesa, California
  - Investigational Site Number 840274, La Mesa, California
  - Investigational Site Number 840222, Long Beach, California
  - Investigational Site Number 840243, Palm Springs, California
  - Investigational Site Number 840250, Spring Valley, California
  - Investigational Site Number 840209, Temecula, California
  - Investigational Site Number 840297, Torrance, California
  - Investigational Site Number 840272, Tustin, California
  - Investigational Site Number 840223, Walnut Creek, California
  - Investigational Site Number 840249, Colorado Springs, Colorado
  - Investigational Site Number 840331, Denver, Colorado
  - Investigational Site Number 840299, Boca Raton, Florida
  - Investigational Site Number 840285, Boynton Beach, Florida
  - Investigational Site Number 840221, Bradenton, Florida
  - Investigational Site Number 840233, Clearwater, Florida
  - Investigational Site Number 840212, Coral Gables, Florida
  - Investigational Site Number 840266, Coral Gables, Florida
  - Investigational Site Number 840204, Hialeah, Florida
  - Investigational Site Number 840248, Hollywood, Florida
  - Investigational Site Number 840226, Jacksonville, Florida
  - Investigational Site Number 840318, Jacksonville, Florida
  - Investigational Site Number 840224, Jacksonville, Florida
  - Investigational Site Number 840228, Miami, Florida
  - Investigational Site Number 840238, Miami, Florida
  - Investigational Site Number 840302, Miami, Florida
  - Investigational Site Number 840337, Miami Beach, Florida
  - Investigational Site Number 840227, New Port Richey, Florida
  - Investigational Site Number 840303, North Miami Beach, Florida
  - Investigational Site Number 840225, Ocala, Florida
  - Investigational Site Number 840291, Orlando, Florida
  - Investigational Site Number 840316, Orlando, Florida
  - Investigational Site Number 840216, Oviedo, Florida
  - Investigational Site Number 840332, Palm Harbor, Florida
  - Investigational Site Number 840288, Pembroke Pines, Florida
  - Investigational Site Number 840325, Port Charlotte, Florida
  - Investigational Site Number 840309, St. Petersburg, Florida
  - Investigational Site Number 840251, Tampa, Florida
  - Investigational Site Number 840339, West Palm Beach, Florida
  - Investigational Site Number 840245, Atlanta, Georgia
  - Investigational Site Number 840323, Stockbridge, Georgia
  - Investigational Site Number 840236, Honolulu, Hawaii
  - Investigational Site Number 840283, Idaho Falls, Idaho
  - Investigational Site Number 840278, Chicago, Illinois
  - Investigational Site Number 840320, Chicago, Illinois
  - Investigational Site Number 840276, Springfield, Illinois
  - Investigational Site Number 840314, Avon, Indiana
  - Investigational Site Number 840317, Avon, Indiana
  - Investigational Site Number 840214, Des Moines, Iowa
  - Investigational Site Number 840232, Overland Park, Kansas
  - Investigational Site Number 840287, Topeka, Kansas
  - Investigational Site Number 840344, Lexington, Kentucky
  - Investigational Site Number 840231, Murray, Kentucky
  - Investigational Site Number 840348, Metairie, Louisiana
  - Investigational Site Number 840290, New Orleans, Louisiana
  - Investigational Site Number 840208, Baltimore, Maryland
  - Investigational Site Number 840301, Rockville, Maryland
  - Investigational Site Number 840289, Fall River, Massachusetts
  - Investigational Site Number 840253, Haverhill, Massachusetts
  - Investigational Site Number 840270, Madison Heights, Michigan
  - Investigational Site Number 840300, Omaha, Nebraska
  - Investigational Site Number 840210, Omaha, Nebraska
  - Investigational Site Number 840263, Omaha, Nebraska
  - Investigational Site Number 840349, Las Vegas, Nevada
  - Investigational Site Number 840201, Las Vegas, Nevada
  - Investigational Site Number 840256, Las Vegas, Nevada
  - Investigational Site Number 840306, Hamilton, New Jersey
  - Investigational Site Number 840203, Sea Girt, New Jersey
  - Investigational Site Number 840295, Sicklerville, New Jersey
  - Investigational Site Number 840269, Albuquerque, New Mexico
  - Investigational Site Number 840310, New Hyde Park, New York
  - Investigational Site Number 840247, Asheville, North Carolina
  - Investigational Site Number 840296, Greensboro, North Carolina
  - Investigational Site Number 840275, Morganton, North Carolina
  - Investigational Site Number 840330, Cleveland, Ohio
  - Investigational Site Number 840307, Columbus, Ohio
  - Investigational Site Number 840229, Norman, Oklahoma
  - Investigational Site Number 840219, Bend, Oregon
  - Investigational Site Number 840240, Philadelphia, Pennsylvania
  - Investigational Site Number 840308, Tipton, Pennsylvania
  - Investigational Site Number 840252, Greer, South Carolina
  - Investigational Site Number 840237, Spartanburg, South Carolina
  - Investigational Site Number 840294, Dakota Dunes, South Dakota
  - Investigational Site Number 840260, Bristol, Tennessee
  - Investigational Site Number 840262, Chattanooga, Tennessee
  - Investigational Site Number 840342, Corpus Christi, Texas
  - Investigational Site Number 840268, Dallas, Texas
  - Investigational Site Number 840292, Dallas, Texas
  - Investigational Site Number 840315, Dallas, Texas
  - Investigational Site Number 840242, Dallas, Texas
  - Investigational Site Number 840326, Edinburg, Texas
  - Investigational Site Number 840338, Houston, Texas
  - Investigational Site Number 840218, Houston, Texas
  - Investigational Site Number 840328, Houston, Texas
  - Investigational Site Number 840259, Houston, Texas
  - Investigational Site Number 840327, Pearland, Texas
  - Investigational Site Number 840282, San Antonio, Texas
  - Investigational Site Number 840202, Murray, Utah
  - Investigational Site Number 840343, Salt Lake City, Utah
  - Investigational Site Number 840239, Burke, Virginia
  - Investigational Site Number 840206, Manassas, Virginia
  - Investigational Site Number 840246, Renton, Washington
  - Investigational Site Number 840311, Milwaukee, Wisconsin
- Bulgaria (5):
  - Investigational Site Number 100205, Blagoevgrad
  - Investigational Site Number 100203, Byala
  - Investigational Site Number 100201, Plovdiv
  - Investigational Site Number 100204, Plovdiv
  - Investigational Site Number 100206, Sofia
- Canada (12):
  - Investigational Site Number 124204, Brampton
  - Investigational Site Number 124211, Etobicoke
  - Investigational Site Number 124208, Laval
  - Investigational Site Number 124214, London
  - Investigational Site Number 124210, Montreal
  - Investigational Site Number 124218, Montreal
  - Investigational Site Number 124206, Pointe-Claire
  - Investigational Site Number 124216, Saint-Laurent
  - Investigational Site Number 124219, Sherbrooke
  - Investigational Site Number 124201, Thornhill
  - Investigational Site Number 124209, Thornhill
  - Investigational Site Number 124212, Toronto
- Czechia (5):
  - Investigational Site Number 203201, Brno
  - Investigational Site Number 203205, Brno
  - Investigational Site Number 203204, Havířov
  - Investigational Site Number 203203, Prague
  - Investigational Site Number 203202, Prague
- Denmark (9):
  - Investigational Site Number 208205, Aalborg
  - Investigational Site Number 208203, Esbjerg
  - Investigational Site Number 208209, Hellerup
  - Investigational Site Number 208202, Herlev
  - Investigational Site Number 208206, Hvidovre
  - Investigational Site Number 208210, Kolding
  - Investigational Site Number 208207, København NV
  - Investigational Site Number 208201, Odense C
  - Investigational Site Number 208204, Viborg
- Estonia (3):
  - Investigational Site Number 233204, Tallinn
  - Investigational Site Number 233203, Tartu
  - Investigational Site Number 233205, Tartu
- Finland (5):
  - Investigational Site Number 246208, Helsinki
  - Investigational Site Number 246202, Kokkola
  - Investigational Site Number 246207, Oulu
  - Investigational Site Number 246206, Tampere
  - Investigational Site Number 246205, Turku
- Hungary (6):
  - Investigational Site Number 348205, Balassagyarmat
  - Investigational Site Number 348201, Budapest
  - Investigational Site Number 348207, Budapest
  - Investigational Site Number 348212, Budapest
  - Investigational Site Number 348210, Budapest
  - Investigational Site Number 348202, Úrhida
- Japan (12):
  - Investigational Site Number 392214, Fujimi
  - Investigational Site Number 392215, Fujimi
  - Investigational Site Number 392206, Ise-Shi
  - Investigational Site Number 392217, Kitaazumi-Gun
  - Investigational Site Number 392208, Matsumoto
  - Investigational Site Number 392210, Matsumoto-Shi
  - Investigational Site Number 392205, Midori
  - Investigational Site Number 392203, Mito
  - Investigational Site Number 392216, Sakai
  - Investigational Site Number 392213, Shimotsuke
  - Investigational Site Number 392218, Shunan-Shi
  - Investigational Site Number 392204, Yamagata
- Latvia (5):
  - Investigational Site Number 428206, Riga
  - Investigational Site Number 428203, Riga
  - Investigational Site Number 428205, Riga
  - Investigational Site Number 428202, Sigulda
  - Investigational Site Number 428201, Ventspils
- Lithuania (5):
  - Investigational Site Number 440203, Kaunas
  - Investigational Site Number 440204, Kaunas
  - Investigational Site Number 440201, Klaipėda
  - Investigational Site Number 440202, Klaipėda
  - Investigational Site Number 440205, Vilnius
- Netherlands (6):
  - Investigational Site Number 528204, Almere Stad
  - Investigational Site Number 528209, Beek
  - Investigational Site Number 528205, Breda
  - Investigational Site Number 528207, Leiderdorp
  - Investigational Site Number 528203, Rotterdam
  - Investigational Site Number 528202, Velp
- Puerto Rico (6):
  - Investigational Site Number 840709, Cagua
  - Investigational Site Number 840706, Carolina
  - Investigational Site Number 840704, San Juan
  - Investigational Site Number 840710, San Juan
  - Investigational Site Number 840703, San Juan
  - Investigational Site Number 840708, San Juan
- Romania (11):
  - Investigational Site Number 642208, Bacau
  - Investigational Site Number 642212, Bucharest
  - Investigational Site Number 642201, Bucharest
  - Investigational Site Number 642202, Cluj-Napoca
  - Investigational Site Number 642213, Oradea
  - Investigational Site Number 642207, Reşiţa
  - Investigational Site Number 642205, Sibiu
  - Investigational Site Number 642203, Târgu Mureş
  - Investigational Site Number 642204, Târgu Mureş
  - Investigational Site Number 642206, Timișoara
  - Investigational Site Number 642209, Timișoara
- Slovakia (6):
  - Investigational Site Number 703205, Banská Bystrica
  - Investigational Site Number 703202, Bardejov
  - Investigational Site Number 703203, Bratislava
  - Investigational Site Number 703201, Levice
  - Investigational Site Number 703206, Levice
  - Investigational Site Number 703207, Lučenec
- Sweden (4):
  - Investigational Site Number 752205, Kristianstad
  - Investigational Site Number 752206, Malmo
  - Investigational Site Number 752201, Stockholm
  - Investigational Site Number 752204, Vällingby

REFERENCES:
- [Result] Bolli GB, Riddle MC, Bergenstal RM, Ziemen M, Sestakauskas K, Goyeau H, Home PD; on behalf of the EDITION 3 study investigators. New insulin glargine 300 U/ml compared with glargine 100 U/ml in insulin-naive people with type 2 diabetes on oral glucose-lowering drugs: a randomized controlled trial (EDITION 3). Diabetes Obes Metab. 2015 Apr;17(4):386-94. doi: 10.1111/dom.12438. Epub 2015 Feb 12. PMID 25641260
- [Derived] Yale JF, Aroda VR, Charbonnel B, Sinclair AJ, Trescoli C, Cahn A, Bigot G, Merino-Trigo A, Brulle-Wohlhueter C, Bolli GB, Ritzel R. Glycaemic control and hypoglycaemia risk with insulin glargine 300 U/mL versus glargine 100 U/mL: A patient-level meta-analysis examining older and younger adults with type 2 diabetes. Diabetes Metab. 2020 Apr;46(2):110-118. doi: 10.1016/j.diabet.2018.10.002. Epub 2018 Oct 23. PMID 30366067
- [Derived] Bolli GB, Wysham C, Fisher M, Chevalier S, Cali AMG, Leroy B, Riddle MC. A post-hoc pooled analysis to evaluate the risk of hypoglycaemia with insulin glargine 300 U/mL (Gla-300) versus 100 U/mL (Gla-100) over wider nocturnal windows in individuals with type 2 diabetes on a basal-only insulin regimen. Diabetes Obes Metab. 2019 Feb;21(2):402-407. doi: 10.1111/dom.13515. Epub 2018 Oct 2. PMID 30160030
- [Derived] Yale JF, Pettus JH, Brito-Sanfiel M, Lavalle-Gonzalez F, Merino-Trigo A, Stella P, Chevalier S, Buzzetti R. The effect of concomitant DPPIVi use on glycaemic control and hypoglycaemia with insulin glargine 300 U/mL (Gla-300) versus insulin glargine 100 U/mL (Gla-100) in people with type 2 diabetes: A patient-level meta-analysis of EDITION 2 and 3. PLoS One. 2018 Jan 25;13(1):e0190579. doi: 10.1371/journal.pone.0190579. eCollection 2018. PMID 29370218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1396 participants were screened, of whom 518 participants were screen failure and 878 participants were randomized.
Groups:
- HOE901-U300: HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily (evening) for 12 months in combination with non-insulin antihyperglycemic drug(s).
- Lantus (Insulin Glargine): Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily (evening) for 12 months in combination with non-insulin antihyperglycemic drug(s).
Period: Overall Study
Arm/Group | HOE901-U300 | Lantus (Insulin Glargine)
Started | 439 | 439
Treated | 435 | 438
Modified Intent-To-Treat Population | 432 (Participants who received at least 1 dose of drug, had both baseline, at least 1 post-baseline data) | 430 (Participants who received at least 1 dose of drug, had both baseline, at least 1 post-baseline data)
Completed | 337 | 314
Not Completed | 102 | 125
Not completed — Randomized But Not Treated | 4 | 1
Not completed — Adverse Event | 10 | 8
Not completed — Lack of Efficacy | 2 | 5
Not completed — Protocol Violation | 11 | 12
Not completed — Received Rescue Therapy | 14 | 22
Not completed — Personal Reason | 34 | 45
Not completed — Lost to Follow-up | 11 | 18
Not completed — Selection Criterion/Protocol Violation | 9 | 9
Not completed — Site Closure/Site Withdrawal | 1 | 4
Not completed — Perceived Lack of Efficacy | 3 | 1
Not completed — Non Serious Hypoglycemia | 2 | 0
Not completed — No More Need of Insulin | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population: all screened participants (who originally met inclusion criteria and signed informed consent) allocated to a treatment group and recorded in Interactive Voice/Web Response System (IVRS/IWRS) database, regardless of whether treatment was used or not. Participants were analyzed in treatment group to which they were randomized.
Groups:
- HOE901-U300: HOE901-U300 SC injection once daily for 12 months in combination with non-insulin antihyperglycemic drug(s).
- Lantus: Lantus SC injection once daily for 12 months in combination with non-insulin antihyperglycemic drug(s).
- Total: Total of all reporting groups
Arm/Group | HOE901-U300 | Lantus | Total
Number analyzed (Participants) | 439 | 439 | 878
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (9.9) | 57.2 (10.3) | 57.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 185 | 371
  Male | 253 | 254 | 507
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 32.8 (6.9) | 33.2 (6.6) | 33.0 (6.7)
Duration of Diabetes [Mean (Standard Deviation); unit: years] — Number of participants analyzed for this baseline characteristics = 435 and 436 in HOE901-U300 and Lantus arm, respectively.
  years | 10.11 (6.49) | 9.57 (6.22) | 9.84 (6.36)
Basal Insulin Daily Dose [Mean (Standard Deviation); unit: units per kilogram (U/kg)] — Number of participants analyzed for this baseline characteristics = 432 and 436 in HOE901-U300 and Lantus arm, respectively.
  units per kilogram (U/kg) | 0.193 (0.027) | 0.193 (0.034) | 0.193 (0.031)
Glycated Hemoglobin A1c (HbA1c) [Number; unit: participants]
  Less Than (<) 8% | 141 | 142 | 283
  Greater Than or Equal to (>=) 8% | 298 | 297 | 595

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Month 6 Endpoint
Description: Only HbA1c measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 Endpoint is either the observed value at Month 6 visit or value retrieved according to time windows.
Time Frame: Baseline, Month 6
Population: Modified Intent-to-Treat (mITT) population:randomized participants who received at least 1 dose, had baseline and at least 1 post-baseline data of any efficacy variable, irrespective of compliance. Number of participants analyzed=participants included in mITT population with baseline and at least 1 post-baseline HbA1c data (Week 12 and/or Month 6).
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 402 | 394
percentage of hemoglobin | -1.42 (0.047) | -1.46 (0.048)
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Analysis was performed using mixed model for repeated measurements (MMRM) with treatment groups, strata of screening HbA1c (<8.0, >=8.0%), geographical region (Non-Japan; Japan), visit and visit-by-treatment groups interaction as fixed categorical effects; baseline HbA1c and baseline HbA1c-by-visit interaction as continuous fixed covariates; Test type: Non-Inferiority or Equivalence — Stepwise closed testing approach was used to assess non-inferiority and superiority sequentially: 1. Non-inferiority of HOE901-U300 vs Lantus: Upper bound of two-sided 95% confidence interval (CI) of difference between HOE901-U300 and Lantus on mITT population is <0.4%. 2. Superiority (only if non-inferiority has been demonstrated): Upper bound of two-sided 95% CI for difference in mean change in HbA1c from baseline to endpoint between HOE901-U300 and Lantus on mITT population is <0; Least Squares (LS) Mean Difference = 0.04, 95% CI 2-sided [-0.090 to 0.174], Standard Error of Mean 0.067

2. Secondary Outcome: Percentage of Participants With At Least One Severe and/or Confirmed Nocturnal Hypoglycemia From Start of Week 9 to Month 6
Description: Nocturnal hypoglycemia was hypoglycemia that occurred between 00:00 and 05:59 hours (clock time), regardless the participant was awake or woke up because of the event. Severe hypoglycemia was an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Confirmed hypoglycemia was an event associated with plasma glucose less than or equal to (<=) 3.9 millimoles per liter (mmol/L) (70 milligram per deciliter [mg/dL]). Only nocturnal hypoglycemia occurring before initiation of rescue therapy were considered in the analysis. Week 9 and Month 6 value correspond to the observed value at Week 9 and Month 6 visit respectively.
Time Frame: Week 9 Up to Month 6
Population: Modified intent-to-treat population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 432 | 430
percentage of participants | 15.5 | 17.4
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; A one-sided test (at alpha=0.025) for superiority of HOE901-U300 over Lantus was to be performed in case the non-inferiority of HOE901-U300 vs Lantus for the primary endpoint was demonstrated. Analysis was performed using Cochran-Mantel-Haenszel (CMH) method stratified by randomization strata of screening HbA1c (<8.0, >=8.0%), randomization strata of geographical region (Non-Japan; Japan); Test type: Superiority or Other; p = 0.4536, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.66 to 1.20]

3. Secondary Outcome: Change in Preinjection Self-Monitored Plasma Glucose (SMPG) From Baseline to Month 6 Endpoint
Description: Pre-injection SMPG was measured within 30 minutes prior to the injection of the study drug. Except for baseline value average of preinjection SMPG was assessed by the mean of at least 3 SMPG calculated over the 7 days preceding the assessment visit. Only preinjection SMPG measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 Endpoint is either the observed value at Month 6 visit or value retrieved according to time windows.
Time Frame: Baseline, Month 6
Population: mITT population. Number of participants analyzed = participants included in the mITT population with baseline and at least one pre-injection SMPG assessment (Week 2, Week 4, Week 8, Week 12, Month 4 and/or Month 6)
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 207 | 222
mmol/L | -2.16 (0.162) | -2.33 (0.156)
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Change in pre-injection SMPG was analyzed using MMRM model with treatment groups, strata of screening HbA1c (<8.0, >=8.0%), geographical region (Non-Japan; Japan), visit and visit-by-treatment groups interaction as fixed categorical effects; baseline preinjection SMPG value and baseline preinjection SMPG value-by-visit interaction as continuous fixed covariates; Test type: Superiority or Other; LS Mean Difference = 0.17, 95% CI 2-sided [-0.275 to 0.605], Standard Error of Mean 0.224

4. Secondary Outcome: Variability of Preinjection SMPG at Month 6 Endpoint
Description: Pre-injection SMPG was measured within 30 minutes prior to the injection of the study drug. Variability was assessed by the mean of coefficient of variation calculated as 100 multiplied by (standard deviation/mean) over at least 3 SMPG measured during the 7 days preceding the assessment visit. Only preinjection SMPG measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 Endpoint is either the observed value at Month 6 visit or value retrieved according to time windows.
Time Frame: Month 6
Population: mITT population. Number of participants analyzed = participants included in the mITT Population with at least one pre-injection SMPG variability assessment (Week 2, Week 4, Week 8, Week 12, Month 4 and/or Month 6).
Measure: Least Squares Mean (Standard Error); unit: percentage of mean
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 422 | 418
percentage of mean | 18.70 (0.502) | 18.33 (0.521)

5. Secondary Outcome: Percentage of Participants With HbA1c <7% at Month 6
Description: Only HbA1c measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 value corresponds to the observed value at Month 6 visit.
Time Frame: Month 6
Population: mITT Population. Participants without any available Month 6 HbA1C assessment were considered as failures (non-responders).
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 432 | 430
percentage of participants | 43.1 | 42.1

6. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Month 6 Endpoint
Description: Only FPG measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 Endpoint is either the observed value at Month 6 visit or value retrieved according to time windows.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants included in the mITT population with baseline and at least one post-baseline FPG assessment (Week 12 and/or Month 6).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 398 | 387
mmol/L | -3.41 (0.103) | -3.80 (0.105)

7. Secondary Outcome: Percentage of Participants With FPG <5.6 mmol/L (100 mg/dL) at Month 6
Description: Only FPG measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 value corresponds to the observed value at Month 6 visit.
Time Frame: Month 6
Population: mITT Population. Participants without any available FPG assessment at Month 6 were considered as failures (non-responders).
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 432 | 430
percentage of participants | 26.2 | 29.5

8. Secondary Outcome: Change in 8-Point SMPG Profiles Per Time Point From Baseline to Month 6
Description: Change in each time-point of 8-point SMPG profile: 03:00 hours (clock time) at night; before and 2 hours after breakfast; before and 2 hours after lunch; before and 2 hours after dinner; and at bedtime. Only 8-point SMPG profiles measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 value corresponds to the observed value at Month 6 visit.
Time Frame: Baseline, Month 6
Population: mITT Population. Only participants from the mITT population with a value at baseline and at specified timepoint were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 432 | 430
mmol/L
  03:00 at Night Plasma Glucose (n=281,277) | -2.63 (3.24) | -3.01 (3.75)
  Pre-Breakfast Plasma Glucose (n=292,286) | -3.28 (2.72) | -3.72 (2.96)
  2 Hours After Breakfast Plasma Glucose (n=278,278) | -3.69 (3.65) | -4.08 (4.03)
  Pre-Lunch Plasma Glucose (n=289,281) | -2.58 (3.39) | -3.39 (3.76)
  2 Hours After Lunch Plasma Glucose (n=280,269) | -2.19 (3.88) | -3.13 (3.77)
  Pre-Dinner Plasma Glucose (n=291,285) | -2.57 (3.49) | -2.43 (3.79)
  2 Hours After Dinner Plasma Glucose (n=282,269) | -2.36 (3.89) | -2.33 (4.03)
  Bedtime Plasma Glucose (n=249,249) | -2.19 (3.75) | -2.26 (3.66)

9. Secondary Outcome: Change in 24-hour Average 8-point SMPG Profile From Baseline to Month 6 Endpoint
Description: Change in 24-hour average of 8-point SMPG profile. 8-point SMPG was assessed at: 03:00 hours (clock time) at night; before and 2 hours after breakfast; before and 2 hours after lunch; before and 2 hours after dinner; and at bedtime. Only 24-hour average 8-point SMPG measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 Endpoint is either the observed value at Month 6 visit or value retrieved according to time windows.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants included in the mITT population with baseline and at least one post-baseline 24-hour average 8-point SMPG assessment (Week 2, Week 4, Week 8, Week 12, Month 4 and/or Month 6).
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Groups:
- HOE901-U300: HOE901-U300 SC injection once daily for 12 months on top of non-insulin antihyperglycemic drug(s).
- Lantus: Lantus SC injection once daily for 12 months on top of non-insulin antihyperglycemic drug(s).
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 381 | 393
mmol/L | -2.72 (0.088) | -2.90 (0.089)

10. Secondary Outcome: Change in Variability of 24 Hour Average 8-point SMPG Profiles From Baseline to Month 6 Endpoint
Description: Variability is assessed by the mean of coefficient of variation calculated as 100 multiplied by (standard deviation/mean) over at least 5 measurements of the 8-point profiles. Only variability of 24-hour 8-point SMPG measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 Endpoint is either the observed value at Month 6 visit or value retrieved according to time windows.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants included in the mITT population with baseline and at least one post-baseline variability of 24-hour average 8-point SMPG assessment (Week 2, Week 4, Week 8, Week 12, Month 4 and/or Month 6).
Measure: Least Squares Mean (Standard Error); unit: percentage of mean
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 381 | 393
percentage of mean | 1.53 (0.643) | 1.41 (0.647)

11. Secondary Outcome: Change in Daily Basal Insulin Dose From Baseline to Month 6
Description: Only insulin dose measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 value corresponds to the observed value at Month 6 visit.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants included in the mITT population with Baseline and Month 6 basal insulin dose assessment.
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 362 | 340
U/kg | 0.43 (0.29) | 0.34 (0.24)

12. Secondary Outcome: Change in Total Treatment Satisfaction Score Using The Diabetes Treatment Satisfaction Questionnaire (DTSQs) From Baseline to Month 6 Endpoint
Description: DTSQ is a validated measure to assess how satisfied participants with diabetes are with their treatment and how they perceive hyper- and hypoglycemia. It consists of 8 questions which are answered on a Likert scale from 0 to 6. DTSQ treatment satisfaction score is the sum of question 1 and 4-8 scores and ranges between 0 and 36, where higher scores indicate more treatment satisfaction. Only DTSQ total score measurements performed before initiation of rescue therapy were considered in the analysis. Month 6 Endpoint is either the observed value at Month 6 visit or value retrieved according to time windows.
Time Frame: Baseline, Month 6
Population: mITT Population. Number of participants analyzed = participants included in the mITT population with Baseline and at least one post-baseline DTSQ assessment (Week 12 and/or Month 6).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 371 | 367
units on a scale | 4.89 (0.246) | 5.12 (0.251)

13. Secondary Outcome: Percentage of Participants With Hypoglycemia (All and Nocturnal) Events From Baseline up to Month 12
Description: Hypoglycemia events were Severe hypoglycemia (an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions); Documented symptomatic hypoglycemia (typical symptoms of hypoglycemia with plasma glucose level of <=3.9 mmol/L [70 mg/dL]); Asymptomatic hypoglycemia (no typical symptoms of hypoglycemia but plasma glucose level <=3.9 mmol/L); Probable symptomatic hypoglycemia (an event during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination, but was presumably caused by a plasma glucose level <=3.9 mmol/L, symptoms treated with oral carbohydrate without a test of plasma glucose); Relative hypoglycemia (an event during which the person with diabetes reported any of the typical symptoms of hypoglycemia, and interpreted the symptoms as indicative of hypoglycemia, but plasma glucose level >3.9 mmol/L); Severe and/or confirmed a hypoglycemia (plasma glucose <=3.9 mmol/L).
Time Frame: Up to 12 months
Population: Safety population: all participants randomized and exposed to at least one dose of study drug, regardless of the amount of treatment administered. In the event of participants having received treatments different from those assigned according to the randomization schedule, safety analyses were conducted according to treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 435 | 438
percentage of participants
  Any Hypoglycemia Event: All Hypoglycemia | 58.9 | 63.2
  Severe Hypoglycemia: All Hypoglycemia | 1.4 | 2.1
  Documented Symptomatic: All Hypoglycemia | 39.1 | 44.1
  Asymptomatic: All Hypoglycemia | 41.6 | 46.8
  Probable Symptomatic: All Hypoglycemia | 3.2 | 3.0
  Relative: All Hypoglycemia | 10.6 | 11.6
  Severe and/or Confirmed: All Hypoglycemia | 56.3 | 61.2
  Any Hypoglycemia Event: Nocturnal Hypoglycemia | 27.6 | 30.1
  Severe Hypoglycemia: Nocturnal Hypoglycemia | 0.0 | 0.7
  Documented Symptomatic: Nocturnal Hypoglycemia | 18.6 | 20.8
  Asymptomatic: Nocturnal Hypoglycemia | 13.3 | 16.0
  Probable Symptomatic: Nocturnal Hypoglycemia | 0.7 | 0.0
  Relative: Nocturnal Hypoglycemia | 4.4 | 3.2
  Severe and/or Confirmed: Nocturnal Hypoglycemia | 25.3 | 29.5

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of informed consent form up to study completion regardless of seriousness or relationship to study drug.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from first injection of study drug up to 2 day after the last injection of study drug). Analysis was done on safety population.
Arm/Group | HOE901-U300 | Lantus
Serious Adverse Events (participants affected / at risk) | 35/435 | 39/438
Other Adverse Events (participants affected / at risk) | 115/435 | 107/438
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=435) | Lantus (N=438)
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 1
Cataract (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Medical device removal (Surgical and medical procedures) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=435) | Lantus (N=438)
Nasopharyngitis (Infections and infestations) | 41 | 47
Sinusitis (Infections and infestations) | 11 | 23
Upper respiratory tract infection (Infections and infestations) | 45 | 34
Headache (Nervous system disorders) | 36 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.